CLINICAL TRIAL: NCT06540755
Title: Analysis of Pregnancy-Associated Plasma Protein-A and Interleukin-6 Gene Polymorphisms in Patients With Periodontitis
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2022.1611; TDH-2023-10969 (Other: Marmara University Scientific Research Projects Unit (BAPSİS))
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Periodontitis; Polymorphism, Restriction Fragment Length
Keywords: Polymorphism; Pregnancy-Associated Plasma Protein-A; Interleukin-6; genetic
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- H Group: periodontally healthy individuals
  Interventions: Genetic: genetic polymorphism analysis
- P Group: stage 3 grade B and C periodontitis patients
  Interventions: Genetic: genetic polymorphism analysis

INTERVENTIONS:
Genetic: genetic polymorphism analysis — Genotype for IL-6 rs1800795 and PAPP-A rs7020782 polymorphisms were determined using real-time polymerase chain reaction with allele-specific probes.

SUMMARY:
The aim of this study is to evaluate the relationship between pregnancy associated plasma protein-A (PAPP-A) and interleukin-6 (IL-6) gene polymorphisms and stage 3 grade B and C (S3GBC) periodontitis, and to compare periodontitis patients with healthy individuals.

DETAILED DESCRIPTION:
A total of 226 systemically healthy subjects, consisted of 112 S3GBC periodontitis patients (P group) and 114 periodontally healthy individuals (H group) were included in our study. Clinical and demographic data were recorded. Genomic deoxyribonucleic acid (DNA) molecules were obtained from peripheral blood. Genotype for IL-6 rs1800795 and PAPP-A rs7020782 polymorphisms were determined using real-time polymerase chain reaction with allele-specific probes. The genotypic or allelic distributions of PAPP-A and IL-6 gene polymorphisms were similar between groups (p>0.05). Our finding suggests that there is no relationship between PAPP-A and IL-6 gene polymorphismS and S3GBC periodontitis, furthermore no difference was detected between periodontitis patients and healthy individuals regarding this gene polymorphism.

ELIGIBILITY:
Inclusion Criteria:

Participants were eligible for inclusion if they were; systemically healthy non-smokers had not undergone periodontal treatment in the past 6 months had not used antibiotics or anti-inflammatory drugs in the preceding 3 months had not used any medication that could affect periodontal tissues in the past 6 months were 18 years of age or older were not pregnant, and were not lactating.

Exclusion Criteria:

The samples taken cannot be stored under appropriate conditions and are damaged.

The onset of a systemic disease in a systemically healthy individual.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group H: The periodontally healthy individuals had an absence of detectable bone and attachment loss, less than 10% of sites with bleeding on probing, and probing depths of ≤3 mm.
  Group P: Stage III grade B or grade C periodontitis patients were diagnosed on the base of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions
Sampling Method: Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2024-01-28 (Actual)

PRIMARY OUTCOMES:
The genotypic or allelic distributions of PAPP-A and IL-6 gene polymorphisms | baseline
  they were similar between groups

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Dental Faculty Periodontology Departmen, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided